CLINICAL TRIAL: NCT06076590
Title: Impact of Multiple Electrolytes Injection Ⅱ and Saline on Hyperchloremia in Patients With Aneurysmal Subarachnoid Hemorrhage:a Pilot Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2023-035-02
Record Dates: First submitted 2023-09-19; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage; Hyperchloremia
Keywords: saline; balanced crystalloids
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multiple electrolytes solution group (Experimental): Experimental group drugs: Multiple Electrolytes Injection(II) Manufacturer: B.Braun Melsungen AG Dosage Form: Liquid Specification: 500ml/ bag Ingredients: Per 1000ml contains: sodium chloride 6.799g, potassium chloride 0.2984g, calcium chloride 0.3675g, magnesium chloride 0.2033g, sodium acetate 3.266g, L-malic acid 0.671, sodium hydroxide 0.200g Duration :36 months Storage conditions: airtight storage, storage temperature shall not exceed 25, can not be refrigerated or frozen
  Interventions: Drug: maintenance fluid
- saline group (Active Comparator): Control group drug: Sodium chloride injection Manufacturer: Hua Run Shuang He Pharmaceutical Co., LTD. Dosage Form: Liquid Specification: 500ml:4.5g Ingredients: Per 1000ml contains sodium chloride 9.0g Duration: 36 months Storage conditions: airtight storage
  Interventions: Drug: maintenance fluid

INTERVENTIONS:
Drug: maintenance fluid — Patients are randomized to receive ether Multiple electrolytes injection II or Normal Saline for maintenance fluid during the 72 hours after enrollment. Resuscitation fluids and fluids used for drug delivery are not limited.

SUMMARY:
The goal of this pilot randomized trial is to compare the effect of Multiple Electrolytes Injection Ⅱand saline on the occurrence of hyperchloremia within 72h of randomization in patients with aneurysmal subarachnoid hemorrhage(aSAH). A secondary aim was to provide data for the design and power of a large-scale, multicenter, randomized controlled trial.

DETAILED DESCRIPTION:
Background:

The isotonic solutions commonly used in ICUs are saline (0.9% sodium chloride) and balanced crystalloid solutions (Ringer's solution, multiple electrolytes injection, etc.). Studies have shown that the lower chloride in balanced crystalloids compared to saline may result in lower risks of hyperchloremia, acute kidney injury and poor clinical outcome in critical ill patients. As a balanced crystalloid, few evidence was found on multiple electrolytes solution II in patients with aneurysmal subarachnoid hemorrhage (aSAH).

Purpose This study aimed to evaluate the security and feasibility of the study. Moreover, compare the impact of multiple electrolytes injection and saline solution on hyperchloremia in aSAH patients.

Method As a pilot trial of a prospective randomized controlled study, patients with aneurysmal subarachnoid hemorrhage randomly assigned to receive saline or multiple electrolytes injection II as maintenance fluid for 3 days during ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients with aneurysmal subarachnoid hemorrhage;
* Expected ICU stay > 24 hours.

Exclusion Criteria:

* Under 18 years of age;
* Pregnancy;
* Patients at imminent risk for death within 24 hours;
* Patients with a known history of serious cardiovascular, respiratory, kidney, liver, blood, or immune disease;
* Azotemia (BUN > 200μmol/L), hypokalemia (blood potassium < 2.5mmol/L), hypocalcemia (blood calcium < 1.8mmol/L);
* Patients routinely receiving renal replacement therapy (RRT);
* Declined to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Hyperchloremia | At 0 hours, 24 hours, 48 hours, 72 hours after enrollment
  The incidence of hyperchloremia

SECONDARY OUTCOMES:
Hyperchloremia acidosis | At 0 hours, 24 hours, 48 hours, 72 hours after enrollment
  Incidence of hyperchloremia acidosis
AKI | recorded at 24 hours, 48 hours, 72 hours after enrollment
  Incidence of acute kidney injury
RRT | recorded at 24 hours, 48 hours, 72 hours after enrollment
  Incidence of new renal replacement therapy
hospital length of stay | recorded at discharge or 28 days after enrollment
  hospital length of stay
hospitalization expense | recorded at discharge or 28 days after enrollment
  money spend during this hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Jian-Xin, MD, Principal Investigator — Capital Medical University
Locations (1):
- ICU, Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No